CLINICAL TRIAL: NCT03908736
Title: Thinking Zinc: A Study of Zinc Supplementation to Ameliorate Adverse Effects of Mine Waste Exposure on the Navajo Nation
Brief Title: Thinking Zinc: a Study of Zinc Supplements on the Navajo Nation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-381
Record Dates: First submitted 2019-04-01; First posted 2019-04-09 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: DNA Damage; Immune System Disorder
MeSH Terms: conditions — Immune System Diseases | interventions — picolinic acid

STUDY DESIGN:
Intervention Model Description: This is a one-armed cohort intervention of zinc supplementation. Data will be collected for each participant before and after zinc supplementation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm cohort (Other): Baseline experimental measurements will be collected for each individual participant twice prior to zinc supplementation (0 month and 3 month time points). After zinc supplementation, experimental measurements will be collected for each individual participant at the 6 month and 9 month time points. The zinc intervention is zinc picolinate 15 mg once per day for 6 months.
  Interventions: Drug: Zinc Picolinate 15 Mg

INTERVENTIONS:
Drug: Zinc Picolinate 15 Mg — zinc picolinate, 15 mg/day for 6 months

SUMMARY:
This is a study to assess the effect of dietary zinc supplementation to mitigate biomarkers of metal toxicity in exposed tribal populations.

DETAILED DESCRIPTION:
Communities living in proximity to abandoned uranium mines have documented exposures to metals in drinking water, soil and dust. Exposure to these metals, principally uranium and arsenic, and metal mixtures is associated with dysregulation of immune function and other health effects. The objective of this study is to conduct an intervention trial to assess the effect of dietary zinc supplementation to mitigate the toxicity of metal exposures. The current project is part of a larger research effort funded by the NIH Superfund Program to study environmental metals exposures in tribal communities in New Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 21 and 64 years of age
* Lives in or near the participating communities of Blue Gap-Tachee Arizona or Red Water Pond Road Community New Mexico
* Willing to provide blood and urine samples
* Willing to attend study visits on scheduled dates
* Willing to take a daily zinc supplement

Exclusion Criteria:

* Women who are pregnant or nursing or women who plan to become pregnant during the course of the study.
* Individuals who have self-reported diabetes, report that they are undergoing treatment for diabetes, or are currently taking medication for diabetes.
* Known or suspected allergy to zinc.
* Individuals previously diagnosed with syndromes of copper homeostasis (Menkes disease or Wilsons disease).
* Individuals consuming zinc supplements or multivitamins and are unwilling to stop for the duration of the study.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Metal biomonitoring to compare change from baseline versus zinc supplement | Visit 1 (0 months-baseline 1), Visit 2 (3 months-baseline 2), Visit 3 (6 months-zinc 1), Visit 4 (9 months-zinc 2)
  urinary and serum metal levels to be measured by inductively coupled plasma mass spectrometry
Lymphocyte phenotyping to compare change from baseline versus zinc supplement | Visit 1 (0 months-baseline 1), Visit 2 (3 months-baseline 2), Visit 3 (6 months-zinc 1), Visit 4 (9 months-zinc 2)
  Lymphocyte phenotypes will be measured in blood samples
Cytokine level measurement to compare change from baseline versus zinc supplement | Visit 1 (0 months-baseline 1), Visit 2 (3 months-baseline 2), Visit 3 (6 months-zinc 1), Visit 4 (9 months-zinc 2)
  A cytokine panel will be used to measure levels of multiple cytokines in blood samples
Autoantibody measurement to compare change from baseline versus zinc supplement | Visit 1 (0 months-baseline 1), Visit 2 (3 months-baseline 2), Visit 3 (6 months-zinc 1), Visit 4 (9 months-zinc 2)
  Autoantibody panel titers will be measured in blood samples

SECONDARY OUTCOMES:
DNA damage assays to compare change from baseline versus zinc supplement | Visit 1 (0 months-baseline 1), Visit 2 (3 months-baseline 2), Visit 3 (6 months-zinc 1), Visit 4 (9 months-zinc 2)
  DNA damage measurements in cells retrieved from blood samples
PARP activity assays to compare change from baseline versus zinc supplement | Visit 1 (0 months-baseline 1), Visit 2 (3 months-baseline 2), Visit 3 (6 months-zinc 1), Visit 4 (9 months-zinc 2)
  Activity measurement of the DNA repair enzyme poly (ADP ribose) polymerase (PARP)

OTHER OUTCOMES:
Exploratory outcome dietary nutritional intake | Visit 2 (3 months), Visit 4 (9 months)
  Food frequency questionnaire for other nutritional factors that may have impact on immune and/or DNA damage parameters

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers unless the other researchers request and receive specific permission for data from the Navajo Nation Human Research Review Board.